CLINICAL TRIAL: NCT05972369
Title: Comparing Sensory Nerve Conduction and Quantitative Sensory Testing Thresholds Between Matched Patients With Nonspecific Low Back Pain Categorized as Responders or Non-Responders to Exercise Therapy
Brief Title: Sensory Nerve Function and Exercise Therapy Response in Chronic Low Back Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ahram Canadian University (Other)
Responsible Party: Principal Investigator, Mohamed Magdy ElMeligie, Lecturer of Physical Therapy and Director of Electromyography Lab, Ahram Canadian University
Other Study IDs: 012/0701LBP02
Record Dates: First submitted 2023-07-24; First posted 2023-08-02 (Actual); Last update posted 2023-08-02 (Actual); Status verified 2023-07

CONDITIONS: Chronic Low-back Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exercise Responders: ≥30% improvement in pain with 12 weeks of prescribed exercise
  Interventions: Other: 12-Week Tailored Exercise Intervention
- Exercise Non-responders: <30% improvement in pain with 12 weeks of prescribed exercise
  Interventions: Other: 12-Week Tailored Exercise Intervention

INTERVENTIONS:
Other: 12-Week Tailored Exercise Intervention — 12-week individually tailored exercise therapy program based on patient presentation. Supervised physiotherapy plus home exercise

SUMMARY:
This observational study aims to compare measures of sensory nerve function between chronic low back pain patients matched for baseline pain and disability levels who are then classified as responders or non-responders after completing a 12-week tailored exercise program. Measures collected include sural sensory nerve conduction, quantitative sensory testing for pressure and heat pain thresholds, and psychosocial questionnaires. It is hypothesized that baseline sensory nerve dysfunction may be associated with reduced response to exercise therapy in chronic low back pain.

DETAILED DESCRIPTION:
While exercise is commonly prescribed for chronic nonspecific low back pain (NSLBP), patient responses are variable. Differences in baseline sensory nerve function could plausibly contribute to exercise therapy outcomes. This cross-sectional quantitative observational study will investigate if baseline sensory nerve conduction amplitudes and quantitative sensory testing (QST) pain thresholds differ between matched NSLBP patients later categorized as responders or non-responders to a 12-week standardized exercise regime. A sample of 50 NSLBP participants with matched baseline pain and disability will undergo a tailored 12-week exercise intervention and 6-month follow-up. Blinded assessors will perform post-intervention sensory nerve conduction and QST measures. It is hypothesized that exercise therapy responders will show greater improvements in sensory thresholds correlating with pain relief. Results aim to elucidate neural factors associated with long-term exercise therapy outcomes in chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 20-60 years
* Nonspecific chronic low back pain >3 months
* Baseline pain ≥6/10 and disability ≥40%

Exclusion Criteria:

* Radicular leg pain
* Prior lumbar surgery
* Serious spinal pathology

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Adults with chronic nonspecific low back pain matched for baseline pain and disability levels.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2023-08-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Sural Sensory Nerve Conduction Amplitude | Baseline
  Baseline antidromic sural sensory nerve action potential amplitude (measured in microvolts) assessed through nerve conduction study.

SECONDARY OUTCOMES:
Superficial Peroneal Sensory Nerve Conduction Amplitude | Baseline
  Baseline superficial peroneal sensory nerve action potential amplitude (measured in microvolts) assessed through nerve conduction study.
Pressure Pain Threshold | Baseline
  Pressure pain threshold (measured in kg/cm2) assessed using a pressure algometer at the lower back.
Heat Pain Threshold | Baseline
  Heat pain threshold (measured in °C) assessed using a thermode applied to the calf.

CONTACTS AND LOCATIONS:
Overall Officials: Amal Fawzy, Ph.d, Study Director — Faculty of Physical Therapy, Ahram Canadian University
Locations (1):
- Outpatient clinic of faculty of physical therapy, Ahram Canadian University, Al Ḩayy Ath Thāmin, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No